CLINICAL TRIAL: NCT07312227
Title: A Prospective Longitudinal Observational Cohort Study of Pregnant Women Residing at High Altitude in Bolivia
Status: Not yet recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, PI, Massachusetts General Hospital
Other Study IDs: PregHigh
Record Dates: First submitted 2025-12-03; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Hypertensive Disorder of Pregnancy; Pulmonary Arterial Hypertension; Intrauterine Growth Restriction
MeSH Terms: conditions — Toxemia; Pulmonary Arterial Hypertension; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal urine, blood samples, umbilical cord blood samples, placental tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy pregnant women residing at high altitude: Women with uncomplicated pregnancy.
- Symptomatic pregnant women residing at high altitude: Women with pregnancy complicated by obstetric conditions such as hypertensive disorders of pregnancy. Hospitalized.

SUMMARY:
In this study, the investigators will follow two small cohorts of pregnant women: a cohort of healthy women with uncomplicated pregnancies residing at high altitude, and a hospitalized cohort of symptomatic women with pregnancies complicated by obstetric conditions (e.g., preeclampsia), to characterize differences in cardiopulmonary adaptation and nitric oxide (NO) pathway expression at elevations >3,500 m throughout pregnancy and into the postpartum period. The investigators aim to investigate right-sided cardiac impairment induced by chronic hypobaric hypoxemia, its effects on fetal growth, and the potential contribution of cardiovascular nitric oxide depletion to obstetric complications such as preeclampsia, pulmonary arterial hypertension, and right ventricular dysfunction.

DETAILED DESCRIPTION:
To investigate cardiac impairment, the investigators will perform transthoracic echocardiography in all enrolled pregnant women and infants, with a focus on right-sided cardiac anatomy and function, including pulmonary artery pressures, right ventricular thickness, right ventricular systolic performance, and indices of pulmonary vascular load.

To investigate the effects of hypobaric hypoxia on fetal growth, the investigators will measure intrauterine and post-delivery growth parameters, assess placental weight and histologic features, and correlate these findings with maternal oxygenation status and altitude exposure.

To assess nitric oxide production and consumption, the investigators will quantify nitric oxide-related metabolites (NO metabolomics) in maternal blood, umbilical cord blood, and placental tissue in both cohorts, and correlate these biomarkers with preeclampsia, pulmonary arterial hypertension, and right ventricular dysfunction. The investigators will also assess flow-mediated dilation in symptomatic and asymptomatic participants and relate these measures of endothelial function to pulmonary vascular and obstetric outcomes.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* women delivering at participating hospitals at more than 3500 meters
* signed informed consent

Exclusion Criteria:

* multiple pregnancy
* preexisting cardiopulmonary pathologies (CHD, COPD, CKD, NYHA > III)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The two cohorts will be selected from pregnant women who have lived at an altitude greater than 3500 meters throughout pregnancy and at delivery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Pulmonary artery pressures | Late pregnancy (35 ± 4 weeks gestation) and postpartum (6 ± 0.3 weeks)
  Measurement will be performed by transthoracic echocardiography.
Echographic estimate of fetal weight | Late pregnancy (35 ± 4 weeks gestation)
Nitric oxide metabolites | Late pregnancy (35 ± 4 weeks gestation) and postpartum (6 ± 0.3 weeks) for maternal samples, at delivery (neonatal samples)
  Measurement will be performed with a chemiluminescence assay.
RV remodeling echocardiography parameters | Late pregnancy (35 ± 4 weeks gestation) and postpartum (6 ± 0.3 weeks)
Weight at birth | At delivery

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusetts General Hospital